CLINICAL TRIAL: NCT01654510
Title: A Systems Level Intervention for Unemployed Persons With Social Anxiety
Brief Title: A Systems Level Intervention for Unemployed Persons With Social Anxiety Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Joseph Himle, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00017734
Record Dates: First submitted 2012-05-10; First posted 2012-07-31 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy Group (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy Group
- Vocational Services as Usual Control (Active Comparator): Vocational services typically present in a comprehensive vocational service center.
  Interventions: Other: Vocational Services as Usual

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy Group — This is a cognitive behavioral therapy group designed for homeless, unemployed people utelizing vocational rehabilitation services. The group is administered on a bi-weekly basis for four weeks, totalling eight sessions.
  Arms: Cognitive Behavioral Therapy Group
Other: Vocational Services as Usual
  Arms: Vocational Services as Usual Control

SUMMARY:
The goal of the proposed research is to design and develop a culturally appropriate, vocationally focused, sustainable, cognitive-behavioral intervention for unemployed, economically disadvantaged, urban-dwelling persons whose job attainment efforts have been undermined by the presence of social anxiety disorder.

DETAILED DESCRIPTION:
The goal of the proposed research is to gather information from Jewish Vocational Service consumers and employees about the association between social anxiety disorder and unemployment. A recent nationally representative epidemiological study places the lifetime prevalence of DSM-IV SocAD at 12.1% (Kessler et al., 2005). Social anxiety disorder is associated with notable impairments in social functioning (Kessler, 2003; Stein and Kean, 2000). A large majority of people with social anxiety disorder report significant impairment in occupational functioning (Stein, et al., 2000; Turner et al., 1986). Specific impairments include turning down job offers and promotions (Stein, Torgrud, & Walker, 2000), reduced productivity and job performance (Wittchen, et al., 2000), lowered educational attainment & early school dropout (Stein & Kean, 2000), increased unemployment (Heimberg et al.,1990a), financial dependence (Scheier et al, 1992), and reduced income (Magee et al., 1996). Social anxiety disorder likely interferes with job attainment due to job interview avoidance, excessive anxious arousal during job interviews, and limited social networks to provide job leads. Our longitudinal study of mothers receiving welfare found that the diagnosis of social anxiety disorder was the strongest psychiatric predictor of reliance on welfare for support over time. We have also completed a study that identifies social anxiety disorder as the only psychiatric disorder that significantly interferes with attaining work among individuals who participated in an internationally tested, best-practice, vocational services intervention program. We have begun to screen individuals for the presence of social anxiety at Jewish Vocational Service in Detroit, Michigan, where the primary clientele are economically disadvantaged, African Americans who are seeking work. Our screening efforts confirm the association between suspected social anxiety disorder and unemployment in this population. This project will build upon these findings and will interview JVS consumers and employees to gain more insight and knowledge into the relationship between social anxiety disorder and unemployment. It will also inform future research on the design and development of a culturally appropriate, vocationally focused, sustainable, cognitive-behavioral intervention for unemployed, economically disadvantaged, urban-dwelling persons whose job attainment efforts have been undermined by the presence of social anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* JVS service-seeking adults
* Unemployed
* Score at least four on the MINI-SPIN
* Meet structured interview criteria for Social Anxiety Disorder and other study related inclusion criteria described below.

Exclusion Criteria:

* Substance use dependence within the past 1 month
* Current use of opiates or freebase cocaine
* Chronic neurological disorder; mental retardation
* Current bipolar I disorder
* Medical conditions contraindicating study treatment
* Prominent suicidal/homicidal ideation with imminent risk

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2008-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale | April 2008 - March 2012 (4 years)
  The primary symptom measure for assessing treatment outcome will be the Liebowitz Social Anxiety Scale (LSAS: Liebowitz, 1987). It assesses fear and avoidance of several social interaction and performance situations.

SECONDARY OUTCOMES:
Employment Status | April 2008 - March 2012 (4 years)
  Reported number of paid work hours per week and the reported number of weeks working at least 35 hours per week (full-time) during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Himle, PhD, Principal Investigator — University of Michigan

REFERENCES:
- [Derived] Himle JA, Bybee D, Steinberger E, Laviolette WT, Weaver A, Vlnka S, Golenberg Z, Levine DS, Heimberg RG, O'Donnell LA. Work-related CBT versus vocational services as usual for unemployed persons with social anxiety disorder: A randomized controlled pilot trial. Behav Res Ther. 2014 Dec;63:169-76. doi: 10.1016/j.brat.2014.10.005. Epub 2014 Oct 30. PMID 25461793